CLINICAL TRIAL: NCT04234802
Title: A Multi-Level Approach to Heat-Related Illness Prevention in Agricultural Workers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute for Occupational Safety and Health (NIOSH/CDC) (U.S. Federal Agency)
Responsible Party: Principal Investigator, June Spector, Associate Professor, Environmental and Occupational Health Sciences; Department of Medicine, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00000238; 2U54OH007544-16 (NIH)
Record Dates: First submitted 2020-01-14; First posted 2020-01-21 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Heat Stress Disorders
MeSH Terms: conditions — Heat Stress Disorders

STUDY DESIGN:
Intervention Model Description: The study is a parallel, comparison, group intervention study to evaluate the effectiveness of a multi-level Heat Education and Awareness Tools (HEAT) intervention, consisting of worker training and a supervisor heat awareness application, on reducing adverse heat health effects in agricultural workers across a growing season.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HEAT intervention group (Active Comparator): Workers in the intervention group will receive the HEAT training, and supervisors in the intervention group will receive the HEAT awareness application and training on how to use it.
  Interventions: Other: Heat Education and Awareness Tools
- Comparison group (No Intervention): The comparison group will not be offered HEAT trainings or the HEAT awareness application. They will be offered an alternative training on another topic.

INTERVENTIONS:
Other: Heat Education and Awareness Tools — HEAT training will be delivered to agricultural workers by research staff in this study in the spring. HEAT training uses interactive approaches to engage participants and posters with visuals. Training covers types of heat-related illness and treatments, risk factors, appropriate clothing and hydration, and keeping cool in the home and community. The HEAT awareness application was developed in collaboration with Washington State University's AgWeatherNet Program to notify supervisors signed up for the service about hot weather conditions that might increase the risk for adverse health effects for workers. The HEAT awareness application is designed to allow subscribers to select weather stations of interest and view current heat indices as well as maximum daily heat indices forecasted over the following week. This information is coupled with information about health effects and prevention of adverse heat health effects. Materials are provided in English and Spanish.
  Arms: HEAT intervention group

SUMMARY:
The project's primary aim is to evaluate the effectiveness of a multi-level heat prevention approach in reducing adverse heat health effects in outdoor agricultural workers

The secondary aims are to:

* Test the effectiveness of an individual-level training component designed to reduce adverse heat health effects in outdoor agricultural workers
* Evaluate the effectiveness of a workplace supervisor-level heat awareness application intended to support supervisor decisions to reduce the risk of workers experiencing adverse heat health effects

ELIGIBILITY:
Inclusion Criteria:

* Speak English or Spanish, live in same dwelling and work at same farm for the season, farm where participant works must agree to collaborate

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2019-05-22 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Heat-related Illness Symptoms | Approximately three months
  Heat symptoms will be assessed using a short survey conducted in Spanish or English that includes questions about heat-related illness symptoms experienced over the past week. Participants will select one or more symptoms (or select 'none') from a list.
Heat Strain | Approximately three months
  The body's physiological response to heat stress. Core body temperature (degrees C) will be estimated using personal baseline temperature and continuous heart rate during work shifts on several days.

SECONDARY OUTCOMES:
Pre/post Knowledge Assessment | Approximately three months
  Short set of multiple-choice questions based on key points addressed in the one-hour training on recognition, treatment, and prevention of heat-related illness.
Pre/post Supervisor Survey | Approximately three months
  Short set of interview questions to learn about heat safety practices and utilization of the HEAT awareness application for intervention group

CONTACTS AND LOCATIONS:
Overall Officials: June T Spector, MD, MPH, Principal Investigator — University of Washington
Locations (1):
- Farms (confidential), Yakima, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified IPD will be available upon reasonable request and/or will be available in a publicly accessible data repository. IPD will include general demographic variables and summary physiological measurements.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will be available after primary analyses are completed, approximately 1-2 years after data collection is completed. Data will be available indefinitely.

REFERENCES:
- [Derived] Chavez Santos E, Spector JT, Egbert J, Krenz J, Sampson PD, Palmandez P, Torres E, Blancas M, Carmona J, Jung J, Flunker JC. The effect of the participatory heat education and awareness tools (HEAT) intervention on agricultural worker physiological heat strain: results from a parallel, comparison, group randomized study. BMC Public Health. 2022 Sep 15;22(1):1746. doi: 10.1186/s12889-022-14144-2. PMID 36104813
- [Derived] Marquez D, Krenz JE, Chavez Santos E, Torres E, Palmandez P, Sampson PD, Blancas M, Carmona J, Spector JT. The Effect of Participatory Heat Education on Agricultural Worker Knowledge. J Agromedicine. 2023 Apr;28(2):187-198. doi: 10.1080/1059924X.2022.2058667. Epub 2022 Apr 17. PMID 35345983
- [Derived] Krenz J, Santos EC, Torres E, Palmandez P, Carmona J, Blancas M, Marquez D, Sampson P, Spector JT. The multi-level heat education and awareness tools [HEAT] intervention study for farmworkers: Rationale and methods. Contemp Clin Trials Commun. 2021 Jun 8;22:100795. doi: 10.1016/j.conctc.2021.100795. eCollection 2021 Jun. PMID 34169175